CLINICAL TRIAL: NCT05907759
Title: A Phase II Study of Daratumumab for Relapsed/Refractory Primary Effusion Lymphoma, Plasmablastic Lymphoma, and Multicentric Castleman Disease
Brief Title: Daratumumab for Relapsed/Refractory Primary Effusion Lymphoma, Plasmablastic Lymphoma, and Multicentric Castleman Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10001538; 001538-C
Record Dates: First submitted 2023-06-15; First posted 2023-06-18 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06-26

CONDITIONS: Lymphoma, Primary Effusion
Keywords: Multicentric Castleman Disease; Non-Hodgkin Lymphoma; Kaposi Sarcoma Herpesvirus; HIV; CD38; B cell lymphoproliferative diseases
MeSH Terms: conditions — Lymphoma, Primary Effusion; Multi-centric Castleman's Disease; Lymphoma, Non-Hodgkin; Sarcoma, Kaposi

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Treatment with daratumumab SC
  Interventions: Drug: Daratumumab SC

INTERVENTIONS:
Drug: Daratumumab SC — Daratumumab SC (daratumumab and hyaluronidase) is administered subcutaneously (SC) as 1800 mg/30,000 units weekly for a total of 8 weeks (8 doses) followed by every 2 weeks for a total of 16 weeks (8 doses) followed by every 4 weeks for up to 96 weeks (24 doses)

SUMMARY:
Background:

Primary effusion lymphoma (PEL), plasmablastic lymphoma (PBL), and Multicentric Castleman Disease (MCD) are aggressive forms of cancer that affects cells in the immune system and lymph nodes. How they develop is not well understood, and these diseases do not respond well to standard treatments for other types of lymphomas.

Objective:

To test a drug treatment (daratumumab SC) in people with PEL, PBL, or MCD.

Eligibility:

People aged 18 and older with PEL, PBL, or MCD who must have failed to respond to therapy or they must be unable to receive standard treatment for the disease.

Design:

Participants will be screened. They will have a physical exam with blood tests. They will have imaging scans and tests of their heart and lung function. They may need to have a biopsy: tissue or fluid will be collected. They will have an eye exam.

Daratumumab SC is given as an injection into the fat under the skin in the abdomen. This takes 3 to 5 minutes. Participants will receive the treatment once a week for 8 weeks; then every 2 weeks for 16 weeks; then every 4 weeks for up to 24 months.

Participants will have other tests during the study period. These may include lumbar punctures: A needle will be inserted between the bones of the spine to draw some fluid from the area around the spinal cord. Participants may also have a thoracentesis: A needle or plastic tube will be inserted into the space around the lungs to withdraw fluid. Participants will have more imaging scans and blood tests.

Follow-up visits will continue after treatment ends. Participants will be in the study for up to 5 years.

DETAILED DESCRIPTION:
Background

* Primary effusion lymphoma (PEL) is an aggressive B cell lymphoma caused by the Kaposi sarcoma herpesvirus (KSHV) with clinicopathologic and molecular profiles distinct from other HIV-related lymphomas.
* Plasmablastic lymphoma (PBL) is an aggressive B-cell lymphoma frequently caused by Epstein-Barr virus (EBV) with frequent extranodal presentations involving the bones and gastrointestinal tract.
* Immunophenotypically, PEL and PBL are post-germinal center B cell neoplasms expressing surface markers consistent with plasmacytic differentiation, such as CD45, CD38, CD138, MUM-1, and IRF4, similar to that of multiple myeloma (MM).
* Outcomes for PEL and PBL treated with front-line combination chemotherapy are inferior to those of other HIV-associated lymphomas, and second-line cytotoxic chemotherapy is often ineffective, and profound immunosuppression often prevents this approach.
* In the second-line setting, chemotherapy-sparing treatments that do not contribute to further immune suppression may be more effective. In addition, patients with PEL often have concurrent KS, which can be severely exacerbated by immune suppression and contributes to mortality in PEL.
* Kaposi sarcoma herpesvirus-associated multicentric Castleman disease (KSHV-MCD) is a rare lymphoproliferative disorder that develops predominantly in people with HIV with inflammatory symptoms associated with high levels of interleukin-6 (IL-6), KSHV-encoded viral IL-6 (vIL-6), and other cytokines.
* The pathologic hallmark of KSHV-MCD is the presence of KSHV-infected Lambda-restricted plasmablasts in the mantle zones of lymph nodes which stain brightly for CD45 and CD38 and negative for CD20.
* KSHV-MCD is generally treated with the anti-CD20 monoclonal antibody, rituximab, with the goal to rapidly improve symptoms and eliminate reservoirs of KSHV-infected plasmablasts.
* Concurrent Kaposi sarcoma is often exacerbated by or develops during rituximab therapy and contributes to morbidity in KSHV-MCD.
* Daratumumab is a human monoclonal antibody that binds to a unique region on CD38 and induces killing of CD38-expressing cells via antibody-dependent cell-mediated cytotoxicity (ADCC), complement-dependent cytotoxicity (CDC), and apoptosis.
* Daratumumab also depletes immunosuppressive non-plasma cells that express CD38 thereby reducing local immunosuppression and stimulating an increase in T-helper cells, cytotoxic T cells, T-cell functional response, and T-cell receptor (TCR) clonality in the tumor microenvironment.

Objective

-To evaluate the partial response (PR) plus complete response (CR) rate (further referred to as the overall response rate [ORR]) of daratumumab SC in participants with relapsed/refractory PEL or PBL and/or symptomatic KSHV-MCD or who are ineligible for front-line chemotherapy

Eligibility

* Age >=18 years
* Participants with pathologically confirmed relapsed and/or refractory PEL, including extracavitary variant and KSHV-associated large cell lymphoma, PBL, or ineligible for front line chemotherapy
* Participants with PEL or PBL must have:

  * Measurable or assessable disease
  * Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0-3
  * Received first-line curative-intent therapy for PEL or PBL, unless such therapy is contraindicated
* Participants with KSHV-MCD must have:

  * ECOG PS (PS) 0-3
  * At least one clinical symptom and at least one laboratory abnormality attributable to KSHV-MCD

Design

* This is a Phase 2 study to evaluate the response rate of daratumumab SC in participants with relapsed/refractory PEL or PBL, and/or symptomatic KSHV-MCD.
* The study will accrue up to 12 evaluable participants with PEL or PBL and up to 12 evaluable participants with KSHV-MCD.
* For participants with relapsed/refractory PEL or PBL, daratumumab SC will be administered subcutaneously (SC) as 1800 mg/30,000 units weekly for a total of 8 weeks (8 doses) followed by every 2 weeks for a total of 16 weeks (8 doses) followed by every 4 weeks for up to 96 weeks (24 doses) in the absence of off-treatment criteria.
* For participants with symptomatic KSHV-MCD, daratumumab SC will be administered SC as 1800 mg/30,000 units weekly for 8 weeks. If response assessment indicates progressive or stable disease, daratumumab SC will be given every 2 weeks for 8 additional doses for up to 24 weeks (6 months).

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants must have primary effusion lymphoma (PEL), including extracavitary variant and KSHV-associated large cell lymphoma, plasmablastic lymphoma (PBL), and/or KSHV-associated multicentric Castleman disease pathologically that relapsed and/or is refractory after front-line chemotherapy or be ineligible for front-line chemotherapy
* Age >= 18 years.
* Any HIV status
* Participants with HIV must be receiving or will initiate an effective combination antiretroviral therapy (ART) regimen and must have an undetectable HIV VL which is defined as <200 copies/mL.
* Participants with PEL or PBL must meet the following criteria:

  * Must have measurable or assessable lymphoma
  * ECOG performance status 0-2 or 3 if secondary to PEL or PBL
  * Adequate hematological and renal functions as defined below:

    * Hemoglobin (Hgb) > 7 g/dL
    * Creatinine clearance (CrCl) >= 15 mL/min/1.73 m^2
  * Must have received first-line curative-intent therapy (anthracycline-containing chemotherapy) for PEL or PBL, unless such therapy is contraindicated due to infection that precludes combination chemotherapy (such as progressive multifocal leukoencephalopathy) or if there is a contraindication to receiving CHOP or EPOCH (such as multi-organ failure).
* Participants with KSHV-MCD must meet the following criteria:

  * ECOG performance status 0-2 or 3 if secondary to MCD
  * Adequate hematological and renal functions as defined below:

    * Hemoglobin (Hgb) > 7 g/dL
    * Creatinine clearance (CrCl) >= 15 mL/min/1.73 m^2
  * At least one clinical symptom attributed to KSHV-MCD

    * Fever (>38 degrees Celsius)
    * Fatigue
    * Gastrointestinal symptoms
    * Respiratory/sinus symptoms
    * Rash
  * At least one laboratory abnormality attributed to KSHV-MCD

    * Anemia (Hgb [men] < 12.5 g/dL, Hgb [women] < 11 g/dL)
    * Thrombocytopenia (< 150 K/microL)
    * Hypoalbuminemia (< 3.4 g/dL)
    * Hyponatremia (< 135 mmol/L)
    * Elevated C-reactive protein (CRP) (> 3 mg/L)
* For participants with evidence of chronic hepatitis B virus (HBV) infection, participants must be on suppressive therapy with an undetectable VL.
* Participants who are seropositive for hepatitis C virus (HCV)are eligible only in the setting of a sustained virologic response [SVR], defined as aviremia, at least 12 weeks after completion of antiviral therapy.
* Participants that have received investigational agents on other clinical trials must have had a washout period of 2 weeks or 5 drug half-lives, whichever is longer.
* Women of child-bearing potential (WOCBP) must agree to use an effective (dual) form of contraception (barrier, surgical sterilization, abstinence) prior to study entry and for the duration of study participation and for 3 months after the last dose of study drug. WOCBP must refrain from egg donations during the study and for 3 months after the last dose of daratumumab.
* Men must agree to use an effective method of contraception (barrier, surgical sterilization, abstinence) for the duration of the study treatment and up to 3 months after the last dose of the study drug(s). We also will recommend men with female partners of childbearing potential to ask female partners to be on an effective birth control (hormonal, intrauterine device [IUD], surgical sterilization).
* Breastfeeding participants must be willing to discontinue breastfeeding from study treatment initiation through 3 months after the last dose of the study drug.
* Participants must understand and sign a written informed consent document.

EXCLUSION CRITERIA:

* Participants who have had anticancer treatment within the last 2 weeks unless the cancer treatment is for a malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial, such as local treatment for carcinoma in situ or hormonal therapy for prostate or breast carcinoma. Toxicity related to prior therapies other than hair loss and neuropathy must have resolved to grade 1.
* KS requiring urgent treatment with cytotoxic chemotherapy.
* Bilirubin (total) > 1.5 times the upper limit of normal; aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 3 times the upper limit of normal (ULN);

EXCEPTIONS:

* Total bilirubin >= 5 mg/dL in participants with Gilbert's syndrome as defined by > 80% unconjugated
* If the elevated total bilirubin or AST/ALT are due to ART or lymphoma

  * ANC < 1000/mm^3 and platelets < 75,000/mm^3 unless related to lymphoma and/or KSHV-MCD or prior therapy.
  * No life-threatening or organ-threatening manifestations of KSHV-MCD.
  * Clinically significant cardiac disease, including:
* Myocardial infarction within 6 months of randomization, or an unstable or uncontrolled disease/condition related to or affecting cardiac function (e.g., unstable angina, congestive heart failure, New York Heart Association Class IIIIV).
* Uncontrolled cardiac arrhythmia

  * Chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) < 50% of predicted normal.
  * Moderate or severe persistent asthma within the past 2 years, or uncontrolled asthma of any classification. Note that participants who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed to participate in the study.
  * Pregnant people as evaluated by a positive serum or urine beta-human chorionic gonadotropin (Beta-hCG) test
  * Participants with severe uncontrolled intercurrent illness, evaluated by history, physical exam and chemistry panel. Participants with severe intercurrent illnesses attributed to lymphoma may be eligible per PI s or designee s discretion.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2034-08-01 (Estimated); Study Completion 2035-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | at 9 and 17 weeks, and every 12 weeks from week 25 to the end of therapy
  Percentage of participants with the best overall response of CR or PR to therapy

SECONDARY OUTCOMES:
Safety of daratumumab | From first dose through 30 days after the end of treatment
  Adverse events (AEs) will be reported by type and grade of toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Robert Yarchoan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be shared
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data from this study may be requested from other researchers at least 1 year after the completion of the primary endpoint.
Access Criteria: Data from this study may be requested by contacting the PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001538-C.html